CLINICAL TRIAL: NCT07066540
Title: Open Multicenter Prospective Observational Trial of the Efficacy and Safety of Use of Drug Product Reamberin® Solution for Infusion, 1.5 % (Scientific Technological Pharmaceutical Firm "POLYSAN") for Pathogenetic Therapy of Viral Enteric Infection in Children Aged 1-6 Years Old
Brief Title: Trial of the Efficacy and Safety of Use of Drug Product Reamberin® for Pathogenetic Therapy of Viral Enteric Infection in Children Aged 1-6 Years Old
Status: Recruiting | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: REAMBERIN-05-2022
Record Dates: First submitted 2025-05-13; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Viral Enteric Infection
Keywords: viral enteric infection; reamberin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Reamberin® in daily dose 10 mL/kg + normal saline (NaCl)/5 % or 10 % solution of glucose
  Interventions: Drug: Reamberin® solution for infusion, 1.5 %
- Control group: Normal saline NaCl/Ringer's solution/5 % or 10 % solution of glucose

INTERVENTIONS:
Drug: Reamberin® solution for infusion, 1.5 % — Reamberin® in daily dose 10 mL/kg
  Groups: Treatment group

SUMMARY:
To assess the efficacy and safety of use of drug product Reamberin® solution for infusion, 1.5 % (Scientific Technological Pharmaceutical Firm "POLYSAN") for pathogenetic therapy of viral enteric infection in children aged 1-6 years old in routine clinical practice. Trial population: children of both sexes at the age of 1-6 years old inclusive with viral enteric infection.

ELIGIBILITY:
Inclusion Criteria:

1. Children of both sexes at the age of 1 to 6 years old inclusive;
2. Diagnosis "Viral and other specified intestinal infections" (code according to the International Statistical Classification of Diseases and Related Health Problems 10th Revision(ICD-10): A08),
3. Clinical signs of endogenous intoxication (nausea, vomiting, hyperthermia, headache, muscle pain, asthenia, adynamia, etc.);
4. Indication for parenteral rehydratation (infusion therapy);
5. Decision of a physician on prescribing drug product Reamberin® solution for infusion, 1.5 % (Scientific Technological Pharmaceutical Firm "POLYSAN") in the daily dose of 10 mL/kg and normal saline NaCl/5 % or 10 % solution of glucose or normal saline NaCl/Ringer's solution/5 % or 10 % solution of glucose;
6. To confirm the diagnosis by laboratory tests, biological material was taken;
7. Informed Consent Form on Participation in the Observational Program signed and dated by a parent/legal representative of the patient.

Exclusion Criteria:

1. Individual intolerance or known hypersensitivity to sodium meglumine, sodium succinate, and/or normal saline (NaCl), solution of glucose, Ringer's solution or excipients of drug product Reamberin® based on data of medical history;
2. Contraindications to prescription of drug product Reamberin®;
3. Necessity in surgical interventions during the observational program;
4. Patients previously enrolled in this trial but discontinued participation due to any any reason;
5. Administration of antibiotics or succinate-containing drug products (Cytoflavin, Mexidol, etc.) and solutions containing malate;
6. Other conditions that, according to the Investigator, prevent enrollment of a patient into the observational trial or can result in premature discontinuation of the observational trial by the patient

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children of both sexes at the age of 1-6 years old inclusive with viral enteric infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in groups who continued to receive infusion therapy 24 hours and 48 hours after the start of the treatment | 24 hours, 48 hours
  Share of patients in groups who continued to receive infusion therapy 24 h (Visit 2) and 48 h (Visit 3) after the start of the treatment
Average duration of infusion therapy in groups, expressed in days | Day 10
  Average duration of infusion therapy in groups, expressed in days
Average durations of symptoms of damage of the gastrointestinal tract in groups | Day 10
  Average durations of symptoms of damage of the gastrointestinal tract (nausea, vomiting, diarrhea) in groups, expressed in days;
Average duration of symptoms of intoxication in groups | Day 10
  Average duration of symptoms of intoxication (asthenia, lethargy, hypodynamia) in groups, expressed in days
Share of patients in groups with moderate form and severe form 48 hours after the start of the treatment | 48 hours
  Share of patients in groups with moderate form (11-15 points according to the Vesikari scale) and severe form (16 and more points according to the Vesikari scale) 48 hours after the start of the treatment (Visit 3);
Average duration of stay of patients in an inpatient healthcare facility | Day 10
  Average duration of stay of patients in an inpatient healthcare facility in treatment groups, expressed in days

SECONDARY OUTCOMES:
Average volume of infusion therapy relative to body weight | Day 10
  Average volume of infusion therapy relative to body weight, expressed in milliliters
Dynamics of intoxication symptoms after 24 hours and 48 hours | 24 hours, 48 hours
  Dynamics of intoxication symptoms (weakness, lethargy, hypodynamia), assessed by VAS (Visual analog scale) after 24 hours (Visit 2) and 48 hours (Visit 3) from the start of infusion therapy compared to Visit 1;
Proportion of patients with electrolyte disturbances after 24 hours | 24 hours
  Proportion of patients with electrolyte disturbances after 24 hours (Visit 2) from the start of infusion therapy compared to Visit 1 (among patients who underwent electrolyte level testing at Visits 1 and 2);
Proportion of patients with base deficit (BE) less than 2 mmol/L after 24 hours | 24 hours
  Proportion of patients with base deficit (BE) less than 2 mmol/L after 24 hours from the start of infusion therapy (among patients who underwent this testing at Visits 1 and 2);
Dynamics of fever severity after 24 hours and 48 hours | 24 hours, 48 hours
  Dynamics of fever severity after 24 hours (Visit 2) and 48 hours (Visit 3) from the start of infusion therapy compared to Visit 1, expressed in degrees Celsius;
Average duration of fever | Day 10
  Average duration of fever, expressed in days
Average duration of stay in the ICU | Day 10
  Average duration of stay in the ICU (intensive care unit), expressed in hours (among patients transferred into ICU)
Dynamics of symptoms of damage of the GI tract 24 hours and 48 hours | 24 hours, 48 hours
  Dynamics of symptoms of damage of the GI (gastrointestinal) tract (nausea, vomiting, and diarrhea) 24 hours (Visit 2) and 48 hours (Visit 3) after the start of infusion therapy as compared to Visit 1;
Dynamics of severity of dehydratation according to the CDS clinical scale 24 hours and 48 hours after the start of infusion therapy | 24 hours, 48 hours
  Dynamics of severity of dehydratation according to the CDS (Clinical Dehydration Scale) clinical scale 24 hours (Visit 2) and 48 hours (Visit 3) after the start of infusion therapy as compared to Visit 1, expressed in points;
Dynamics of changes of parameters of complete blood count and leukocytic index of intoxication 24 hours and 48 hours | 24 hours, 48 hours
  Dynamics of changes of parameters of complete blood count and leukocytic index of intoxication 24 hours (Visit 2) and 48 hours (Visit 3) after the start of treatment as compared to Visit 1 (among patients who underwent this analysis).

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (7):
  - South Ural State Medical University, Chelyabinsk
  - Khimki Clinical Hospital, Khimki
  - Kuban State Medical University, Krasnodar
  - Infectious Diseases Clinical Hospital No. 1, Moscow
  - Z.A. Bashlyaeva Children's City Clinical Hospital, Moscow
  - Penza Regional Clinical Center for Specialized Types of Medical Care, Penza
  - Children's Scientific and Clinical Center for Infectious Diseases of the Federal Medical and Biological Agency, Saint Petersburg
- Samarkand State Medical University, Samarkand, Uzbekistan